CLINICAL TRIAL: NCT00333255
Title: Preoperative and Postoperative Nevanac 0.1% Compared to Acular LS for the Treatment of Ocular Inflammation Associated With Cataract Surgery
Brief Title: Nepafenac Opthalmic Suspension 0.1% Compared to Acular LS for Treatment of Inflammation After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-04-41
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Drug: Nepafenac Ophthalmic Suspension, 0.1%

SUMMARY:
The purpose of this study is to compare the effectiveness of Nepafenac Ophthalmic Suspension, 0.1% eye drops to Acular LS eye drops, used before and after cataract surgery, for treating inflammation in the eye.

ELIGIBILITY:
Inclusion Criteria:

* planned cataract extraction with posterior chamber intraocular lens implantation

Exclusion Criteria:

* Under 10

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who are a clinical success at Day 14 postoperative visit (where a "clinical success" is defined as aqueous cells < grade 1 and aqueous flare = grade 0 at the current visit and all subsequent visits).

SECONDARY OUTCOMES:
Percentage of patients who are clinically cured, clinical successes, treatment failure, clinically significant inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Maxwell, Study Director — Study Director
Locations (1):
- Lehmann Eye Center, Nacogdoches, Texas, United States